CLINICAL TRIAL: NCT05865990
Title: Multicenter, Single-arm, 3 Cohort, Phase II Trial of HER3-DXd in Patients With Active Brain Metastases From Metastatic Breast Cancer and Non-small Cell Lung Cancer, and in Patients With Leptomeningeal Disease From Advanced Solid Tumors
Brief Title: HER3-DXd in Breast Cancer and NSCLC Brain Metastases and Solid Tumor Leptomeningeal Disease
Acronym: TUXEDO-3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDOPP575; 2023-503251-10-00 (Other: EU CT number)
Record Dates: First submitted 2023-04-10; First posted 2023-05-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Breast Cancer; Advanced Non-Small Cell Squamous Lung Cancer; Solid Tumor, Adult
Keywords: Brain Metastasis; Leptomeningeal Disease
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Meningeal Neoplasms | interventions — patritumab deruxtecan

STUDY DESIGN:
Intervention Model Description: An international, multicenter, single-arm, three-cohort, two-stage optimal Simon's design, phase II clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patritumab deruxtecan (HER3-DXd) (Experimental): HER3-DXd will be dosed at 5.6 mg/kg body weight as an intravenous (IV) infusion administered on day 1 (D1) of each 21-day cycle for patients from all cohorts until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.
  * Cohort 1: MBC with untreated or progressing BM after local treatment.
  * Cohort 2: aNSCLC with untreated or progressing BM after local treatment.
  * Cohort 3: advanced solid tumor with treatment-naive LMD or LMD progressing after radiotherapy.
  Interventions: Drug: Patritumab deruxtecan

INTERVENTIONS:
Drug: Patritumab deruxtecan — HER3 directed antibody drug conjugate (ADC) that is comprised of a fully human anti-HER3 immunoglobulin gamma-1 (IgG1) monoclonal antibody attached to a topoisomerase I inhibitor payload (an exatecan derivative, DXd) via a stable tetrapeptide-based cleavable linker.
  Other Names: HER3-DXd

SUMMARY:
The goal of this phase II clinical trial] is to analyze the efficacy of patritumab deruxtecan (HER3-DXd) in patients with metastatic breast cancer (MBC) or advanced non-small cell lung cancer (aNSCLC) with active brain metastases (BM) who have received at least one line of systemic therapy in the advanced setting, or patients with active leptomeningeal carcinomatosis/disease (LMD) after radiotherapy from an advanced solid tumor who do not need immediate local treatment, and have not received prior treatment with an anti-HER3 targeted drug].

The main questions it aims to answer are:

* The intracranial objective response rate (ORR-IC) per local investigator as judged by best central nervous system (CNS) response according to Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria of HER3-DXd in patients with active BM from MBC (Cohort 1) and aNSCLC (Cohort 2).
* The overall survival (OS) rate at 3 months of HER3-DXd in patients with advanced solid tumors with untreated LMD (Cohort 3).

Participants will receive HER3-DXd on day (D1) of each 21-day cycle until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.

Researchers will compare historical groups to see if HER3-DXd positively impacts patient outcomes.

DETAILED DESCRIPTION:
In this international, multicenter, single-arm, multicohort, optimal Simon's design phase II clinical trial, patients will be treated with HER3-DXd, which is a new antibody-drug conjugate (ADC) that targets specifically the HER3 protein (which is expressed in the surface of tumor cells) and that is attached to deruxtecan.

Male or female patients ≥ 18 years of age with MBC or aNSCLC with untreated or progressing BM after local treatment, or solid tumor patients with treatment-naive LMD or patients with recurrence of LMD after radiotherapy, and no need for immediate local treatment. All patients except for patients with LMD (cohort 3) must have received one prior line of systemic therapy in the advanced setting.

Note I: prior systemic treatments for breast cancer (BC) eligible patients would be defined as follows:

* triple negative breast cancer (TNBC) patients must have received at least one line of prior systemic therapy for advanced disease.
* luminal BC patients must have received at least one line of endocrine therapy (ET) and one line of chemotherapy (CT) in the advanced setting.
* HER2-positive (HER2[+]) BC patients must have progressed on at least two previous treatments with HER2-targeted therapies in the advanced setting.

Note II: prior systemic treatments for NSCLC eligible patients would be defined as follows:

* Patients without and with epidermal growth factor receptor (EGFR) (and other) activating driver alterations are allowed.
* Patients with activating driver alterations must have received at least one prior line of an approved genotype directed therapy.
* Patients with EGFR T790M mutation following first-line treatment with erlotinib, gefitinib, afatinib, or dacomitinib must have received second-line osimertinib, and have documentation of radiological disease progression on treatment.

After confirmed eligibility, patients will be assigned to one of three study cohorts as follows:

* Cohort 1 (N=20): 10 patients in the stage I and 10 patients in the stage II. MBC with untreated or progressing BM after local treatment.
* Cohort 2 (N=20): 10 patients in the stage I and 10 patients in the stage II. aNSCLC with untreated or progressing BM after local treatment.
* Cohort 3 (N=20): 10 patients in the stage I and 10 patients in the stage II. Advanced solid tumor with treatment-naive LMD or LMD progressing after radiotherapy.

Upon meeting all selection criteria, patients enrolled in the study will receive patritumab deruxtecan (HER3-DXd), which will be dosed at 5.6 mg/kg body weight as an intravenous (IV) infusion administered on day 1 (D1) of each 21-day cycle.

Patients will receive treatment disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.

Patients discontinuing the study treatment period prematurely, will enter a post-treatment follow-up period during which survival and new anti-cancer therapy information will be collected, until end of study (EoS) or study termination, whichever occurs first.

ELIGIBILITY:
* GENERAL INCLUSION CRITERIA (Patients will be included in the study only if they meet all the following inclusion criteria):

  1. Patient must be capable to understand the purpose of the study and have signed written informed consent form (ICF) prior to beginning specific protocol procedures.
  2. Age ≥ 18 years at the time of signing ICF.
  3. Life expectancy ≥ 6 weeks.
  4. Karnofsky Performance Status (KPS) ≥70%, Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
  5. Patient must be able to tolerate therapy.
  6. Availability and willingness to provide the most recently available tumor tissue sample (formalin-fixed and paraffin-embedded [FFPE], no cytology/cell block, no bone/decalcified bone sample) of primary tumor or any metastatic site from biopsy preferably collected after last round of prior treatment and ≤ 6 months prior to HER3-DXd treatment, if possible, at the time of inclusion for retrospective exploratory biomarker testing. If archival tissue is not available, a newly obtained baseline biopsy of an accessible tumor lesion is required prior to start of study treatment (unless not possible because of inaccessible tumor location or safety concerns).
  7. No indication for immediate local therapy.
  8. Patient has adequate bone marrow, liver, and renal function:

     1. Hematological (without platelet, red blood cell transfusion, and/or granulocyte colony-stimulating factor support within 7 days before first study treatment dose): White blood cell (WBC) count > 3.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100.0 x109/L, and hemoglobin ≥ 10.0 g/dL (≥ 6.2 mmol/L).
     2. Hepatic: Serum albumin ≥ 2.5 g/dL; total bilirubin ≤ 1.5 times upper limit of normal (ULN) (≤ 3 in patients with liver metastases or know history of Gilbert's disease); alkaline phosphatase (ALP) ≤ 2.5 times ULN; aspartate transaminase (AST); alanine transaminase (ALT) ≤ 3 times ULN (≤ 5 in patients with liver metastases); international normalized ratio (INR) < 1.5.
     3. Renal: serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min/1.73 m2 based on Cockcroft-Gault glomerular filtration rate estimation for patients with creatinine levels above institutional normal.
  9. Patients must have received at least 1 prior line of systemic treatment* in the advanced setting.

     * Prior systemic treatments for eligible patients with BC are defined as follows:

       * Patients with triple-negative breast cancer (TNBC) must have received at least one line of prior systemic therapy for advanced disease.
       * Patients with luminal BC must have received at least one line of ET and one line of CT in the advanced setting.
       * Patients with HER2-positive BC must have progressed to at least two previous treatments with HER2-targeted therapies in the advanced setting.
     * Prior systemic treatments for eligible patients with aNSCLC are defined as follows:

       * Patients without activating driver alterations must have received at least one prior line of standard of care systemic therapy for locally advanced or metastatic disease.
       * Patients with activating driver alterations must have received at least one prior line of an approved genotype-directed therapy.
       * Patients with EGFR T790M mutation who received first-line treatment with erlotinib, gefitinib, afatinib, or dacomitinib must have received second-line treatment with osimertinib and have documentation of radiological disease progression.
  10. Resolution of all acute toxic effects of prior anti-cancer therapy to grade ≤ 1 as determined by the US National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (v.5.0).

      Note: Except for alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion.
  11. For women of childbearing potential: agreement to remain abstinent (must refrain from heterosexual intercourse) or use highly effective contraceptive methods, or two effective contraceptive methods, as defined in the protocol, during the treatment period and for at least 7 months after the last dose of study treatment, whichever is longer. Women of childbearing potential must have a negative serum pregnancy test within 14 days before study treatment initiation and must agree to refrain from donating eggs during the entire study treatment period and for 7 months after the last administration of the study drug.
  12. For male subjects: being surgically sterile or having agreed to true abstinence (must refrain from heterosexual intercourse) or having female partners willing to agree with true abstinence or use barrier contraceptive measures mentioned above during the entire study treatment period and for 4 months after the last administration of the study drug. Male patients must agree to refrain from donating sperm during the entire study treatment period and for 4 months after the last administration of the study drug.
  13. Patient must be accessible for treatment and follow-up.
* SPECIFIC INCLUSION CRITERION FOR COHORT 1 AND COHORT 2 (Cohort 1 and cohort 2 patients will be included in the study only if they meet all the following inclusion criteria):

  1. Histologically documented BC (cohort 1) or NSCLC of squamous or non-squamous histologic types (cohort 2).
  2. Newly diagnosed BM or BM progressing after local treatment.
  3. Measurable disease according to Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria, with at least one measurable brain lesion of ≥10 mm on T1-weighted, gadolinium-enhanced MRI.
* SPECIFIC INCLUSION CRITERION FOR COHORT 1 AND COHORT 2 (Cohort 1 and cohort 2 patients will be included in the study only if they meet all the following inclusion criteria):

  1. Histologically documented BC (cohort 1) or NSCLC of squamous or non-squamous histologic types (cohort 2).
  2. Radiologically documented metastatic disease. 3. Newly diagnosed BM or BM progressing after local treatment. 4. Measurable disease according to Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria, with at least one measurable brain lesion of ≥10 mm on T1-weighted, gadolinium-enhanced MRI.
* SPECIFIC INCLUSION CRITERION FOR COHORT 1 (Cohort 1 patients will be included in the study only if they meet the following inclusion criterion):

  1. Locally determined HER2 status.
* SPECIFIC INCLUSION CRITERIA FOR COHORT 3 (Cohort 3 patients will be included in the study only if they meet all the following inclusion criteria):

  1. Histologically documented solid tumor of any type.
  2. Type I LMD, defined by positive CSF cytology or leptomeningeal biopsy, or type II LMD, defined by clinical findings and neuroimaging only, according to European Society for Molecular Oncology (ESMO) Standard Operating Procedures (SOPs) for Clinical Practice Guideline (CPG) 2017.
  3. Newly diagnosed LMD or LMD progressing after radiotherapy.
* EXCLUSION CRITERIA (Patients will be excluded from the study if they meet any of the following criteria):

  1. Current participation in another therapeutic clinical trial.
  2. Treatment with approved or investigational cancer therapy within 14 days prior to initiation of study drug.
  3. Patients have a concurrent malignancy or malignancy within five years of study enrollment with the exception of carcinoma in situ of the cervix, non-melanoma skin carcinoma, or stage I uterine cancer. For other cancers considered to have a low risk of recurrence, discussion with the Medical Monitor is required.
  4. Previous systemic therapy with any anti-HER3 directed drug.
  5. Known allergy or hypersensitivity to HER3-DXd or any of the drug components.
  6. Radiotherapy or limited-field palliative radiotherapy within seven days prior to study enrolment, or patients who have not recovered from radiotherapy-related toxicities to baseline or grade ≤ 1 and/or from whom ≥ 25% of the bone marrow has been previously irradiated.
  7. Patients with an active cardiac disease or a history of cardiac dysfunction or conduction abnormalities including any of the following:

     1. Unstable angina pectoris or documented myocardial infarction within 6 months prior to study entry.
     2. Symptomatic pericarditis.
     3. Documented congestive heart failure (CHF) (New York Heart Association [NYHA] Class III-IV).
     4. Left ventricular ejection fraction (LVEF) < 50% as determined by multigated acquisition (MUGA) scan or echocardiogram (ECHO).
     5. Ventricular arrhythmias except for benign premature ventricular contractions.
     6. Other cardiac arrhythmias requiring a pacemaker or not controlled with medication.
     7. Long QT syndrome (QTcF interval > 450 ms).
  8. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e., pulmonary emboli within three months of the study enrolment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion etc.), and any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (i.e., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis etc.), or prior pneumonectomy.
  9. History of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
  10. Pregnant or lactating women.
  11. Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study.
  12. Current known infection with hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antibody [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
  13. Known human immunodeficiency virus (HIV) infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA, CD4-positive cells' count ≥ 350, no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 4 weeks on the same anti-HIV medications (meaning there are no expected further changes in that time to the number or type of antiretroviral drugs in the regimen). If an HIV infection meets the above criteria, monitoring of viral RNA load and CD4-positive cells' count is recommended.
  14. History of a major surgical procedure (defined as requiring general anesthesia) or significant traumatic injury within 21 days prior to randomization, or patients who have not recovered from the side effects of any major surgery.
  15. History of uncontrolled seizures, CNS disorders or serious and/or unstable pre-existing psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs or interfering with subject safety.
  16. Patients requiring concomitant use of chronic systemic (intravenously [IV] or oral) corticosteroids at doses higher than 8 mg dexamethasone per day or other immunosuppressive medications except for managing adverse events (AEs), including immune-related adverse events (irAEs) for patients that received immunotherapy in a previous line; (inhaled steroids or intra articular steroid injections are permitted in this study).

      Note: The use of stable corticosteroid therapy in patients with brain metastases can be discussed with the Medical Monitor.
  17. Patients with known substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
  18. Participants who are unable or unwilling to comply with the requirements of the protocol in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Local determination of intracranial objective response rate (ORR-IC) in cohort 1 and cohort 2. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Rate of patients with complete response (CR) or partial response (PR) determined locally by investigator, using Response Assessment in Neuro-Oncology Brain Metastases (RANO)-BM criteria in cohort 1 and cohort 2.
Efficacy: Overall survival (OS) rate at 3 months in cohort 3. | From baseline up to 3 months
  3-month OS, defined as the rate of patients alive at 3 months after treatment initiation in cohort 3.

SECONDARY OUTCOMES:
Efficacy: Central determination of ORR in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  ORR, defined as the rate of patients with CR or PR determined by central review as per RANO-BM in cohort 1 and cohort 2 and per ESMO-EANO in cohort 3 for intracranial lesions, and per RECIST v.1.1 for extracranial and overall lesions (bicompartmental ORR) in all cohorts.
Efficacy: progression-free survival (PFS) in cohort 1, cohort 2, and cohort 3. | From baseline up to 12 months
  PFS, defined as the period from treatment initiation to the first occurrence of disease progression or death from any cause or treatment discontinuation from any other reason, whichever occurs first, that will be centrally reviewed as per RANO-BM for intracranial lesions in cohort 3 and RECIST v.1.1 for extracranial and overall lesions in all cohorts.
Efficacy: bicompartmental clinical benefit rate (CBR) in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  CBR, defined as the rate of patients with objective response (CR or PR), or stable disease for at least 24 weeks, centrally reviewed as per RANO-BM in cohort 1 and cohort 2 and ESMO-EANO in cohort 3 for intracranial lesions, and RECIST v.1.1 for extracranial and overall lesions (bicompartmental CBR) in all cohorts.
Efficacy: disease control rate (DCR) in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  DCR, defined as the rate of patients with objective response (CR or PR), or stable disease (SD), determined by central review as per RANO-BM in cohort 1 and cohort 2 and ESMO-EANO in cohort 3 for intracranial lesions, and RECIST v.1.1 for extracranial and overall lesions (bicompartmental DCR) in all cohorts.
Efficacy: time to response (TTR) in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  TTR, defined as the period from the treatment initiation to time of the first objective tumor response (tumor shrinkage of ≥ 30%) observed for patients who achieved a CR or PR, centrally reviewed as per RANO-BM in cohort 1 and cohort 2 and ESMO-EANO in cohort 3 for intracranial lesions, and RECIST v.1.1 for extracranial and overall lesions in all cohorts.
Efficacy: duration of response (DoR) in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  DOR, defined as the period from the first occurrence of a documented objective response to disease progression or death from any cause, observed for patients who achieved a CR or PR. It will be centrally reviewed as per RANO-BM in cohort 1 and cohort 2 and ESMO-EANO in cohort 3 for intracranial lesions, and RECIST v.1.1 for extracranial and overall lesions in all cohorts.
Efficacy: best percentage of change in tumor burden in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Best percentage of change in tumor burden centrally reviewed as per RANO-BM in cohort 1 and cohort 2 and ESMO-EANO in cohort 3 for intracranial lesions, and RECIST v.1.1 for extracranial and overall measurable lesions in all cohorts.
Efficacy: overall survival (OS) in cohort 1 and cohort 2. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  OS, defined as the period from treatment initiation to death from any cause or last available follow-up in cohort 1 and cohort 2.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Safety and tolerability of HER3-DXd as per National Cancer Institute Common Terminology Criteria for Adverse Events (AEs) Version 5.0 (NCI-CTCAE v.5.0) in all cohorts.
Patient reported outcomes (PROs) with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-30) of patients in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of overall change from baseline in QoL with the EORTC QLQ-C30 scale to measure cancer patients' physical, psychological and social functions in all cohorts. All scales and single items are transformed into scores ranging from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptomatology.
Effects of the tumor and its function with the European Organization for Research and Treatment of Cancer brain cancer-specific Quality of Life Questionnaire (EORTC QLQ-BN20) of patients in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of overall change from baseline of the effects of brain tumors and its treatment on symptoms, functions and health-related quality of life with the brain specific tool (EORTC QLQ-BN20) in all cohorts. All scales and single items are transformed into scores ranging from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptomatology.
Effects of the tumor and its function using the European Organization for Research and Treatment of Cancer breast cancer-specific Quality of Life Questionnaire (EORTC QoL-BR45) of breast cancer patients in cohort 1. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of overall change from baseline of the effects in QoL of breast cancer patients in cohort 1 with the breast specific tool EORTC QLQ-BR45 scale to measure physical, psychological and social functions. All scales and single items are transformed into scores ranging from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptomatology.
Assessment of overall change from baseline of the effects of the tumor in and its treatment in neurologic function using the Neurologic Assessment in Neuro-Oncology (NANO) scale in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Differences in neurologic assessment in NANO scale in all cohorts. High-scale values represent impaired neurological performances. NANO scale differences (values before and after treatment) below or equal to 0 represent a stable or improved neurological performance and vice versa.

OTHER OUTCOMES:
Efficacy endpoints according to HER3 expression level and tumor type in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of the correlation between HER3 expression level and efficacy of HER3-DXd treatment in all cohorts.
Efficacy endpoints according to the prior administration of treatment with or without an antibody drug conjugate (ADC)-based therapy in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of the relationship between the efficacy of HER3-DXd and prior treatment with or without ADC therapy in all cohorts.
Predictive or prognostic biomarkers in MRI and/or CT scan images according to disease activity status or response to treatment in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of the relationship between MRI and/or CT scan images and patient clinical characteristics or efficacy outcomes in all cohorts.
Predictive or prognostic biomarkers in biosamples according to disease activity status or response to treatment in cohort 1, cohort 2, and cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of the relationship between blood and/or tumor sample-based biomarkers and patient clinical characteristics or efficacy outcomes in all cohorts.
Efficacy endpoints according to TROP2 expression level and tumor type in cohorts 1 and 2. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of the relationship between TROP2 expression level and efficacy of HER3-DXd treatment in cohorts 1 and 2.
Efficacy endpoints according to estrogen receptor (ER) expression level and tumor type in cohort 1. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of the relationship between ER expression level and efficacy of HER3-DXd in cohort 1.
Efficacy endpoints according to progesterone receptor (PgR) expression level in cohort 1. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of the relationship between PgR expression level and efficacy of HER3-DXd in cohort 1.
Efficacy endpoints according to HER2 expression level in cohort 1. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of the relationship between HER2 expression level efficacy of HER3-DXd in cohort 1.
Efficacy endpoints according to the prior administration of treatment with or without tucatinib in HER2[+] breast cancer patients in cohort 1. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of the relationship between the efficacy of HER3-DXd and prior treatment with or without tucatinib in HER2[+] breast cancer patients in cohort 1.
Predictive or prognostic biomarkers in cerebrospinal fluid (CSF) samples according to diseas activity status or response to treatment in patients in cohort 3. | From baseline to the date of first documented progression, death from any cause, or treatment discontinuation from any reason, whichever came first, assessed up to 12 months
  Assessment of the relationship between CSF-based biomarkers and patient clinical characteristics or efficacy outcomes in cohort 3 (only if collected as per local guidelines and clinical routine).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Preusser, MD, Principal Investigator — Medical Oncologist. Head of Clinical Division of Oncology, Medical University of Vienna; Rupert Bartsch, MD, PhD, Principal Investigator — Consultant Hematology and Medical Oncology, Medical University of Vienna
Locations (8):
- Austria (2):
  - Salzburg Cancer research Institute-Center for Clinical Cancer and Immunology Trials, Salzburg
  - Medical University of Vienna, Vienna
- Spain (6):
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Beata María Ana, Madrid
  - Hospital Quirónsalud Sagrado Corazón, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Arnau de Vilanova de Valencia, Valencia

REFERENCES:
- [Derived] Bartsch R, Marhold M, Garde-Noguera J, Gion M, Ruiz-Borrego M, Greil R, Valero M, Llombart-Cussac A, Garcia-Mosquera JJ, Arumi M, Cortes J, Campolier M, Guerrero JA, Slebe F, Martinez-Garcia E, Jimenez-Cortegana C, Vaz-Batista M, Oberndorfer F, Furtner J, Fuereder T, Berghoff AS, Preusser M. Patritumab deruxtecan (HER3-DXd) in patients with active brain metastases of breast cancer (TUXEDO-3): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2025 Nov;26(11):1467-1478. doi: 10.1016/S1470-2045(25)00470-X. PMID 41167215
- [Derived] Fuereder T, Garde-Noguera J, Garcia-Mosquera JJ, Ruiz-Borrego M, Valero M, Llombart-Cussac A, Gion M, Greil R, Arumi M, Campolier M, Guerrero JA, Raimondi G, Mancino M, Jimenez-Cortegana C, Vaz-Batista M, Oberndorfer F, Marhold M, Berghoff AS, Furtner J, Bartsch R, Preusser M. Patritumab deruxtecan (HER3-DXd) in patients with active brain metastases of non-small-cell lung cancer (TUXEDO-3): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2025 Nov;26(11):1454-1466. doi: 10.1016/S1470-2045(25)00465-6. PMID 41167214
- [Derived] Preusser M, Garde-Noguera J, Garcia-Mosquera JJ, Gion M, Greil R, Arumi M, Ruiz-Borrego M, Llombart-Cussac A, Valero M, Cortes J, Campolier M, Guerrero JA, Gonzalez-Alonso P, Jimenez-Cortegana C, Rodriguez-Morato J, Vaz-Batista M, Oberndorfer F, Marhold M, Berghoff AS, Furtner J, Fuereder T, Bartsch R. Patritumab deruxtecan in leptomeningeal metastatic disease of solid tumors: the phase 2 TUXEDO-3 trial. Nat Med. 2025 Aug;31(8):2797-2805. doi: 10.1038/s41591-025-03744-1. Epub 2025 May 30. PMID 40447851